CLINICAL TRIAL: NCT00430612
Title: The PACE-MI Registry Study - Outcomes of Beta-blocker Therapy After Myocardial Infarction (OBTAIN)
Acronym: OBTAIN
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeff Goldberger, Principal Investigator, MD, MBA, Professor of Medicine, Northwestern University
Other Study IDs: 469; U01HL080416 (NIH)
Record Dates: First submitted 2007-01-31; First posted 2007-02-02 (Estimated); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Heart Attack; Beta Blockers; Survival
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All Registry Participants: Non-voluntary registry of consecutive patients diagnosed as having a MI at each study site.

SUMMARY:
The purpose of the PACE-MI (OBTAIN) registry is:

* Analyze beta-blocker dose response effect on outcome over two years
* Explore gender and minority differences in beta-blocker utilization and outcomes.

In patients with Myocardial Infarction (MI) discharged from the hospital, beta-blocker dose will be predictive of survival.

Exploratory analyses: Gender and racial effects-gender and race are, similarly, hypothesized to be predictive of post-MI survival.

The existence of interactions between gender and beta-blocker effect as well as race and beta-blocker effect will also be evaluated.

DETAILED DESCRIPTION:
Methods

All patients admitted to the coronary care areas with an acute myocardial infarction will be entered into the registry. At the time of discharge from the coronary care unit, clinical data will be entered. The registry will include approximately 6800 patients.

As there is no intervention in the registry, the data to be collected are standard for quality assurance purposes and cannot practicably be carried out without waivers of consent and HIPAA authorization, there will be no consent specifically for registry patients at baseline. Systems have been implemented to ensure the registry data will remain confidential. Sites have received IRB approval of waiver of consent and HIPAA for the baseline registry data.

Data to be collected will include demographic (including ethnic and race classifications according to NIH guidelines) data and information regarding the index myocardial infarction. Use of beta-blockers at discharge from the coronary care unit will be documented. In addition, beta-blocker use at hospital discharge will be noted. Data for the registry will be obtained from ER notes, admission notes, cardiac catheterization lab reports, medication lists, lab reports, and discharge summaries.

Follow-Up

Follow-up for registry patients will be conducted at year 1 and year 2 post-myocardial infarction. Data may be obtained via medical chart review, phone contact, and Social Security Death Index (SSDI). For follow-up information obtained via chart review or the SSDI, a detailed justification for waiver of HIPAA and consent requirements is attached to this protocol. If phone contact is required with the patient, we are suggesting the following process:

* A letter should be sent out to the patient approximately one week prior to the contact in which the rationale for the study will be provided, as well as a delineation of the patient's right to participate or not to participate (by either providing or not providing the requested information).
* At telephone contact with the patient, the coordinator will document whether the patient consents to provide the information. If the patient consents, the coordinator will proceed to obtain the requested information.
* In the event that the participating institution's IRB requires a written, signed consent for this verbal contact, a written consent form template is provided.

Data collected at follow-up interview will include vital status, beta-blocker use, other cardiac medications and any cardiovascular hospitalizations.

ELIGIBILITY:
Inclusion Criteria

1. Consecutive patients admitted with a myocardial infarction documented by both of the following:

1. cardiac enzymes (CPK elevation > two times or troponin elevation > three times the upper limit of normal for the lab)
2. Electrocardiographic changes and/or symptoms consistent with myocardial infarction (i.e. chest pain, shortness of breath)

No Exclusion Criteria

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non-voluntary registry of consecutive patients diagnosed as having a MI at each study site
Sampling Method: Non-Probability Sample
Enrollment: 7057 (Actual)
Dates: Start 2009-05; Primary Completion 2013-12 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Total mortality at 2 years post myocardial infarction | Measured at Years 1 and 2
  Compare Kaplan Meier survival curves for the following 5 beta-blocker dose groups:
  No beta-blockers - 12.5% (>0 - 12.5%) 25% (>12.5 - 25%) - 50% (>25 - 50%) Full Dose (>50%)

SECONDARY OUTCOMES:
Total mortality - secondary analysis | Measured at Year 1 and Year 2
  Compare Kaplan-Meier survival curves for the following 2 beta-blocker dose groups:
  Very Low Dose (>0-25%) vs. High Dose (≥50%)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Goldberger, MD, MBA, Principal Investigator — Northwestern University
Locations (23):
- United States (22):
  - Little Rock Cardiology Clinic, Little Rock, Arkansas
  - MemorialCare Heart and Vascular Institute - Long Beach Memorial Medical Center, Long Beach, California
  - West Los Angeles VA Medical Center, Los Angeles, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Clarian Health/Methodist Research Institute, Indianapolis, Indiana
  - Henry Ford Hospital, Detroit, Michigan
  - Park Nicollet, Saint Louis Park, Minnesota
  - Winthrop University Hospital, Bethpage, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Strong Memorial Hospital (University of Rochester School of Medicine), Rochester, New York
  - OhioHealth Research Institute, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Amarillo Heart Clinic Research Institute, Inc., Amarillo, Texas
  - Austin Heart PLLC, Austin, Texas
  - Providence Health Center, Waco, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Background] Wikstrand J, Hjalmarson A, Waagstein F, Fagerberg B, Goldstein S, Kjekshus J, Wedel H; MERIT-HF Study Group. Dose of metoprolol CR/XL and clinical outcomes in patients with heart failure: analysis of the experience in metoprolol CR/XL randomized intervention trial in chronic heart failure (MERIT-HF). J Am Coll Cardiol. 2002 Aug 7;40(3):491-8. doi: 10.1016/s0735-1097(02)01970-8. PMID 12142116
- [Background] Metra M, Torp-Pedersen C, Swedberg K, Cleland JG, Di Lenarda A, Komajda M, Remme WJ, Lutiger B, Scherhag A, Lukas MA, Charlesworth A, Poole-Wilson PA. Influence of heart rate, blood pressure, and beta-blocker dose on outcome and the differences in outcome between carvedilol and metoprolol tartrate in patients with chronic heart failure: results from the COMET trial. Eur Heart J. 2005 Nov;26(21):2259-68. doi: 10.1093/eurheartj/ehi386. Epub 2005 Jul 21. PMID 16040619
- [Background] Dobre D, van Veldhuisen DJ, Mordenti G, Vintila M, Haaijer-Ruskamp FM, Coats AJ, Poole-Wilson PA, Flather MD; SENIORS Investigators. Tolerability and dose-related effects of nebivolol in elderly patients with heart failure: data from the Study of the Effects of Nebivolol Intervention on Outcomes and Rehospitalisation in Seniors with Heart Failure (SENIORS) trial. Am Heart J. 2007 Jul;154(1):109-15. doi: 10.1016/j.ahj.2007.03.025. PMID 17584562
- [Background] Cucherat M. Quantitative relationship between resting heart rate reduction and magnitude of clinical benefits in post-myocardial infarction: a meta-regression of randomized clinical trials. Eur Heart J. 2007 Dec;28(24):3012-9. doi: 10.1093/eurheartj/ehm489. Epub 2007 Nov 2. PMID 17981830
- [Background] Kjekshus JK. Importance of heart rate in determining beta-blocker efficacy in acute and long-term acute myocardial infarction intervention trials. Am J Cardiol. 1986 Apr 25;57(12):43F-49F. doi: 10.1016/0002-9149(86)90888-x. PMID 2871745
- [Background] Chen ZM, Pan HC, Chen YP, Peto R, Collins R, Jiang LX, Xie JX, Liu LS; COMMIT (ClOpidogrel and Metoprolol in Myocardial Infarction Trial) collaborative group. Early intravenous then oral metoprolol in 45,852 patients with acute myocardial infarction: randomised placebo-controlled trial. Lancet. 2005 Nov 5;366(9497):1622-32. doi: 10.1016/S0140-6736(05)67661-1. PMID 16271643
- [Background] POISE Study Group; Devereaux PJ, Yang H, Yusuf S, Guyatt G, Leslie K, Villar JC, Xavier D, Chrolavicius S, Greenspan L, Pogue J, Pais P, Liu L, Xu S, Malaga G, Avezum A, Chan M, Montori VM, Jacka M, Choi P. Effects of extended-release metoprolol succinate in patients undergoing non-cardiac surgery (POISE trial): a randomised controlled trial. Lancet. 2008 May 31;371(9627):1839-47. doi: 10.1016/S0140-6736(08)60601-7. Epub 2008 May 12. PMID 18479744
- [Background] Gottlieb S, Harpaz D, Shotan A, Boyko V, Leor J, Cohen M, Mandelzweig L, Mazouz B, Stern S, Behar S. Sex differences in management and outcome after acute myocardial infarction in the 1990s: A prospective observational community-based study. Israeli Thrombolytic Survey Group. Circulation. 2000 Nov 14;102(20):2484-90. doi: 10.1161/01.cir.102.20.2484. PMID 11076821
- [Background] Wilkinson P, Laji K, Ranjadayalan K, Parsons L, Timmis AD. Acute myocardial infarction in women: survival analysis in first six months. BMJ. 1994 Sep 3;309(6954):566-9. doi: 10.1136/bmj.309.6954.566. PMID 7916229
- [Background] Mahon NG, McKenna CJ, Codd MB, O'Rorke C, McCann HA, Sugrue DD. Gender differences in the management and outcome of acute myocardial infarction in unselected patients in the thrombolytic era. Am J Cardiol. 2000 Apr 15;85(8):921-6. doi: 10.1016/s0002-9149(99)00902-9. PMID 10760327
- [Background] Vaccarino V, Krumholz HM, Yarzebski J, Gore JM, Goldberg RJ. Sex differences in 2-year mortality after hospital discharge for myocardial infarction. Ann Intern Med. 2001 Feb 6;134(3):173-81. doi: 10.7326/0003-4819-134-3-200102060-00007. PMID 11177329
- [Background] A randomized trial of propranolol in patients with acute myocardial infarction. I. Mortality results. JAMA. 1982 Mar 26;247(12):1707-14. doi: 10.1001/jama.1982.03320370021023. PMID 7038157
- [Background] Olsson G, Wikstrand J, Warnold I, Manger Cats V, McBoyle D, Herlitz J, Hjalmarson A, Sonneblick EH. Metoprolol-induced reduction in postinfarction mortality: pooled results from five double-blind randomized trials. Eur Heart J. 1992 Jan;13(1):28-32. doi: 10.1093/oxfordjournals.eurheartj.a060043. PMID 1533587
- [Background] Rochon PA, Anderson GM, Tu JV, Clark JP, Gurwitz JH, Szalai JP, Lau P. Use of beta-blocker therapy in older patients after acute myocardial infarction in Ontario. CMAJ. 1999 Nov 30;161(11):1403-8. PMID 10906894
- [Background] Soumerai SB, McLaughlin TJ, Spiegelman D, Hertzmark E, Thibault G, Goldman L. Adverse outcomes of underuse of beta-blockers in elderly survivors of acute myocardial infarction. JAMA. 1997 Jan 8;277(2):115-21. PMID 8990335
- [Background] Gottlieb SS, McCarter RJ, Vogel RA. Effect of beta-blockade on mortality among high-risk and low-risk patients after myocardial infarction. N Engl J Med. 1998 Aug 20;339(8):489-97. doi: 10.1056/NEJM199808203390801. PMID 9709041
- [Background] Haywood LJ. Coronary heart disease mortality/morbidity and risk in blacks. I: Clinical manifestations and diagnostic criteria: the experience with the Beta Blocker Heart Attack Trial. Am Heart J. 1984 Sep;108(3 Pt 2):787-93. doi: 10.1016/0002-8703(84)90672-0. PMID 6148005
- [Background] Hjalmarson A, Elmfeldt D, Herlitz J, Holmberg S, Malek I, Nyberg G, Ryden L, Swedberg K, Vedin A, Waagstein F, Waldenstrom A, Waldenstrom J, Wedel H, Wilhelmsen L, Wilhelmsson C. Effect on mortality of metoprolol in acute myocardial infarction. A double-blind randomised trial. Lancet. 1981 Oct 17;2(8251):823-7. doi: 10.1016/s0140-6736(81)91101-6. PMID 6116950
- [Background] Norwegian Multicenter Study Group. Timolol-induced reduction in mortality and reinfarction in patients surviving acute myocardial infarction. N Engl J Med. 1981 Apr 2;304(14):801-7. doi: 10.1056/NEJM198104023041401. PMID 7010157
- [Background] Viskin S, Kitzis I, Lev E, Zak Z, Heller K, Villa Y, Zajarias A, Laniado S, Belhassen B. Treatment with beta-adrenergic blocking agents after myocardial infarction: from randomized trials to clinical practice. J Am Coll Cardiol. 1995 May;25(6):1327-32. doi: 10.1016/0735-1097(94)00552-2. PMID 7722129
- [Background] The Cardiac Insufficiency Bisoprolol Study II (CIBIS-II): a randomised trial. Lancet. 1999 Jan 2;353(9146):9-13. PMID 10023943
- [Background] Dargie HJ. Effect of carvedilol on outcome after myocardial infarction in patients with left-ventricular dysfunction: the CAPRICORN randomised trial. Lancet. 2001 May 5;357(9266):1385-90. doi: 10.1016/s0140-6736(00)04560-8. PMID 11356434
- [Background] Metoprolol in acute myocardial infarction (MIAMI). A randomised placebo-controlled international trial. The MIAMI Trial Research Group. Eur Heart J. 1985 Mar;6(3):199-226. PMID 2863148
- [Background] American Heart Association. Heart disease and stroke statistics-2009 update. Dallas: American Heart Association; 2009.
- [Background] Dmitrienko A, Molenberghs G, Chuang-Stein C, Offen W. Analysis of clinical trials using SAS: A practical guide. Cary, NC: SAS Institute Inc.; 2005.
- [Background] Westfall PH. Multiple comparisons and multiple tests : using the SAS system. 1. print. ed. Cary NC: SAS Inst.; 1999.
- [Background] Tu JV, Willison DJ, Silver FL, Fang J, Richards JA, Laupacis A, Kapral MK; Investigators in the Registry of the Canadian Stroke Network. Impracticability of informed consent in the Registry of the Canadian Stroke Network. N Engl J Med. 2004 Apr 1;350(14):1414-21. doi: 10.1056/NEJMsa031697. PMID 15070791
- [Derived] Goldberger JJ, Bonow RO, Cuffe M, Liu L, Rosenberg Y, Shah PK, Smith SC Jr, Subacius H; OBTAIN Investigators. Effect of Beta-Blocker Dose on Survival After Acute Myocardial Infarction. J Am Coll Cardiol. 2015 Sep 29;66(13):1431-41. doi: 10.1016/j.jacc.2015.07.047. PMID 26403339